CLINICAL TRIAL: NCT03351790
Title: Assessing the Quality of Upper Gastrointestinal Endoscopy - Factors That Affect it and Validation of a Bespoke Mucosal Visual Scale
Brief Title: Endoscopy Quality Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sandwell & West Birmingham Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Nigel Trudgill, Consultant Gastroenterologist, Sandwell & West Birmingham Hospitals NHS Trust
Other Study IDs: 15GAST29
Record Dates: First submitted 2017-11-20; First posted 2017-11-24 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All included participants: Patients that complete study questionnaire and have endoscopy recorded.
  Interventions: Other: Questionniare only

INTERVENTIONS:
Other: Questionniare only — A pre-procedure questionnaire will be completed by all participants

SUMMARY:
This study seeks to establish factors that influence the view at endoscopy. To achieve this patients, who have been already booked for endoscopy, will complete a questionnaire prior to their procedure. Demographic and endoscopist factors will also be ascertained.

The view at endoscopy will then be reviewed and scored against a rating scale, which will be validated as a first phase of the study. Factors can then be sought that are associated with a good endoscopic view.

ELIGIBILITY:
Inclusion Criteria:

* Any patient booked for routine OGD

Exclusion Criteria:

* Inpatient endoscopy
* Barretts surveillance endoscopy

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients referred for upper GI endoscopy (OGD)
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2018-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
View seen at endoscopy | Endoscopy will be performed as booked for standard care. This will be the same day as consent.
  This is the quality of view seen at endoscopy based upon a bespoke scale